CLINICAL TRIAL: NCT01510379
Title: Median Nerve Acustimulation Plus Medical Anti-emetic Therapy for Control Post-operative Nausea in Patients Undergoing Foregut Surgery: A Randomized Control Trial
Brief Title: Reletex Versus Standard of Care Therapy for Post-Operative Nausea Control in Patients Undergoing Foregut Surgery
Acronym: Reletex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle A Perry (Other)
Responsible Party: Sponsor-Investigator, Kyle A Perry, Assistant Professor General Surgery 614-293-5815, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011H0236
Record Dates: First submitted 2012-01-05; First posted 2012-01-16 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Nausea and Vomiting Post-foregut Surgery
Keywords: nausea; vomiting; post-operative; foregut surgery
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; Promethazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reletex (Active Comparator): Reletex plus scheduled IV ondansetron 4 mg q 6 hours for a total of 4 doses. Breakthrough nausea will be treated using IV promethazine 25 mg q 6 hours prn during the hospital stay and in elixir at the same dose and frequency after discharge.
  Interventions: Device: Reletex; Drug: IV ondansetron 4 mg q 6 hours for a total of 4 doses; Drug: IV promethazine 25 mg q 6 hours prn; Drug: Elixir promethazine 25 mg q 6 hours prn after discharge
- Control (Other): Scheduled IV ondansetron 4 mg q 6 hours for a total of 4 doses. Breakthrough nausea will be treated using IV promethazine 25 mg q 6 hours prn during the hospital stay and in elixir at the same dose and frequency after discharge.
  Interventions: Device: Reletex; Drug: IV ondansetron 4 mg q 6 hours for a total of 4 doses; Drug: IV promethazine 25 mg q 6 hours prn; Drug: Elixir promethazine 25 mg q 6 hours prn after discharge

INTERVENTIONS:
Device: Reletex — Neurostimulation device for prevention/treatment of post-operative nausea and vomiting, Reletex arm.
Drug: IV ondansetron 4 mg q 6 hours for a total of 4 doses
Drug: IV promethazine 25 mg q 6 hours prn
Drug: Elixir promethazine 25 mg q 6 hours prn after discharge

SUMMARY:
The effect a ReletexTM device has on postoperative nausea and vomiting when used with ondansetron after foregut surgery will be studied. A ReletexTM device is a FDA approved wristwatch-like device that painlessly stimulates a nerve in the wrist and has been shown to decrease nausea and vomiting. The investigators will randomize 100 patients who are having a fundoplication for either gastroesophageal reflux disease (GERD), paraesophageal hernia, or Heller Myotomy for achalasia into two groups. A control group will receive scheduled ondansetron for prevention and treatment of postoperative nausea and vomiting and phenergan as needed. The treatment group will wear a ReletexTM wrist band after surgery for 7 days. These patients will also get scheduled ondansetron and phenergan as needed, like the control group. The investigators will compare nausea, retching, and the amount of supplemental nausea medication used between the two groups. The patients will be provided a diary to document their nausea, retching, and medication use.

The hypothesis of this study is that use of the ReletexTM device will reduce post-operative nausea and vomiting, and will reduce post-operative use of anti-emetic medications in patients who have undergone foregut surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Planned fundoplication
* Willingness to comply with randomization and follow-up protocol
* English speaking

Exclusion Criteria:

* < 18 years of age or > 85
* Chronic nausea requiring medical treatment
* Planned concomitant procedures
* Pacemaker or automatic internal cardiac defibrillator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Perry, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at The Ohio State University Wexner Medical Center over a 1 year period.
Pre-assignment Details: Enrolled participants were not excluded from the trial before assignment to groups.
Period: Overall Study
Arm/Group | Reletex | Control
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Reletex: Reletex plus scheduled ondansetron and phenergan prn
- Control: Scheduled ondansetron plus phenergan prn
- Total: Total of all reporting groups
Arm/Group | Reletex | Control | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 74
  >=65 years | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.22) | 58 (16.16) | 57 (15.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 14 | 17 | 31
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Postoperative Nausea and Vomiting Scores Between Groups Treated With a ReletexTM Device and Those Without the Device.
Description: Post-operative Nausea and Vomiting (PONV) Likert scale, 0-10 (0=no PONV, 10=worst PONV).
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reletex | Control
Number analyzed (Participants) | 49 | 51
units on a scale | 1.81 (2.17) [0 to 10] | 2.03 (2.83) [0 to 10]

2. Secondary Outcome: Quantify the Amounts of Phenergan Used Between the Two Groups.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Reletex | Control
Number analyzed (Participants) | 49 | 51
mg | 42 (75.6) | 57.6 (128.2)

ADVERSE EVENTS:
Arm/Group | Reletex | Control
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes